CLINICAL TRIAL: NCT00414219
Title: Visual Prognosis in Non-Penetrating Corneal Blast Injuries
Status: Completed | Type: Observational
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Other Study IDs: WRAMC WU# 04-23010
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2010-12

CONDITIONS: Corneal Foreign Body Following Blast Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Visual quality of patients with corneal eye injuries — Visual quality of patients with corneal eye injuries

SUMMARY:
The purpose of this study is to assess visual quality of patients with non-penetrating, non-metallic, stable corneal foreign bodies. Visual quality will be assessed by examining visual acuity, wavefront analysis and contrast sensitivity. Drawings, photographs, and confocal microscopy will be used to document clinical examination of the cornea at baseline and on follow-up examinations.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Access to medical care at Walter Reed Army Medical Center
* Age 18 years or older
* Corneal foreign bodies from blast injuries
* Available for evaluation at Walter Reed

Exclusion Criteria:

* Residual, recurrent or active ocular disease in the designated eye as determined by exam and history.
* Penetrating ocular trauma or injury to the posterior segment
* Prior history of ocular surgery
* Any physical or mental impairment that would preclude participation in any of the examinations.
* Any ocular abnormality other than corneal foreign bodies that have any impact on vision (i.e. other abnormalities from trauma such as retinal detachment, corneal laceration, traumatic cataract, or abnormalities unrelated to trauma such as herpes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: US Army patients age 18 years and older prsenting with corneal foreign bodies from non-penetrating ocular blast injuries
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2004-11; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dain Brooks, MD, Principal Investigator — Ophthalmology Service, Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States